CLINICAL TRIAL: NCT01780623
Title: A Randomized Controlled Trial of Light Therapy on Biomarkers, Sleep/Wake Activity, and Quality of Life in Individuals With Post-treatment Cancer-related Fatigue
Brief Title: An Investigation of Light Therapy for Cancer-related Fatigue (The LITE Study)
Acronym: LITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Dr. Tavis S. Campbell, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10003569
Record Dates: First submitted 2013-01-22; First posted 2013-01-31 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
Keywords: fatigue; sleep; quality of life; light; cancer
MeSH Terms: conditions — Neoplasms; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright White Light (Experimental): Bright white light exposure every morning for 30 minutes for 28 consecutive days
  Interventions: Device: Bright white light
- Dim Red Light (Active Comparator): Dim red light exposure every morning for 30 minutes for 28 consecutive days
  Interventions: Device: Dim red light

INTERVENTIONS:
Device: Bright white light
  Other Names: Light box; LiteBook
  Arms: Bright White Light
Device: Dim red light
  Other Names: Light box; LiteBook
  Arms: Dim Red Light

SUMMARY:
Cancer-related fatigue is one of the most common and distressing symptoms associated with a cancer diagnosis.Fatigue related to cancer often appears before a diagnosis, worsens during treatment, and lasts for years after treatment in up to 35% of patients. Despite the long-term effects of cancer-related fatigue, the treatment options available are not always appropriate or helpful for all patients.Light therapy is an effective treatment for other disorders related to fatigue. The purpose of the study is to investigate the role of light therapy on quality of life, sleep patterns, and physical measures of immune function and stress hormones in individuals with post-treatment cancer-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Non metastatic cancer
* At least 3 months post chemotherapy/radiation treatment (hormone treatment ok)
* Meets criteria for cancer-related fatigue

Exclusion Criteria:

* Under 18 years of age
* Presence of a sleep disorder other than insomnia or hypersomnia
* Shift work
* Presence of an Axis-I psychiatric condition
* Presence of a medical condition that may impact levels of fatigue
* Presence of conditions contraindicated to the use of light therapy or photosensitizing medications
* Randomization refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in fatigue symptoms from baseline to post-treatment | Baseline, after each treatment week (each week for 4 weeks), and at week 5

SECONDARY OUTCOMES:
Change in objective measures of sleep using wrist actigraphy from baseline to post-treatment | Baseline (for 7 days), week 5 (for 7 days)
Change in subjective measures of sleep using sleep diaries from baseline to post-treatment | Baseline (for 7 days), week 5 (for 7 days)
Change in Pittsburgh Sleep Quality Index scores from baseline to post-treatment | Baseline, week 5
Change in Profile of Mood States scores from baseline to post-treatment | Baseline, week 5
Change in Functional Assessment of Cancer Therapy (General & Fatigue) scores from baseline to post-treatment | Baseline, week 5
Change in salivary cortisol from baseline to post-treatment | Baseline (for 3 days), week 5 (for 3 days)
Change in inflammatory cytokines from baseline to post-treatment | Baseline, week 5
Change in Insomnia Severity Index scores from baseline to post-treatment | Baseline, week 3, week 5

CONTACTS AND LOCATIONS:
Overall Officials: Tavis S Campbell, PhD, Principal Investigator — University of Calgary
Locations (1):
- Behavioural Medicine Laboratory, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Johnson JA, Subnis U, Carlson LE, Garland SN, Santos-Iglesias P, Piedalue KL, Deleemans JM, Campbell TS. Effects of a light therapy intervention on diurnal salivary cortisol in fatigued cancer survivors: A secondary analysis of a randomized controlled trial. J Psychosom Res. 2020 Dec;139:110266. doi: 10.1016/j.jpsychores.2020.110266. Epub 2020 Oct 6. PMID 33070045